CLINICAL TRIAL: NCT03087383
Title: Identification of Genetic Polymorphisms Related to Propofol Requirement and Recovery Through Genome-wide Association Study (GWAS) in Total Intravenous Anesthesia for Clipping of Unruptured Cerebral Aneurysm in Korean Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0008
Record Dates: First submitted 2017-03-07; First posted 2017-03-22 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Unruptured Cerebral Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood obtained from enrolled patients before surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: In adult patients undergoing propofol based TIVA for clipping of unruptured cerebral aneurysm, investigator will collect data regarding recovery after stopping propofol infusion (time for eye opening and extubation), propofol requirement during anesthesia maintenance, and propofol effect site concentration to achieve bispectral index 40 during anesthesia induction, without doing any interventions. Data collection will be established with just observing and recording values displayed in screens of monitoring devices, and reviewing patient charts.
- Retrospective Cohort: In previous study performed in adult patients undergoing propofol based TIVA for clipping of unruptured cerebral aneurysm (NCT02700126, 4-2015-1195), investigator enrolled patients and collected data regarding recovery after stopping propofol infusion (time for eye opening and extubation), propofol requirement during anesthesia maintenance, and propofol effect site concentration to achieve bispectral index 40 during anesthesia induction, without doing any interventions.

SUMMARY:
In neurosurgical anesthesia, propofol based total intravenous anesthesia (TIVA) is frequently used due to brain relaxation and less effect on electrophysiologic monitoring. Response to propofol can vary between individuals and be associated with clinical factors including age and weight, and genetic polymorphism. Because the importance of rapid recovery in neurosurgery with long operation time is emphasized recently, the choice and dose adjustment of anesthetics should be determined according to clinical and genetic factors. Recently, researches about genetic variations have been performed with single nucleotide polymorphism (SNP). The aim of this study is to find SNPs associated with propofol recovery and response through genome-wide association study (GWAS) in Korean adult population undergoing propofol based TIVA for clipping of unruptured cerebral aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Korean adult population undergoing propofol based TIVA for clipping of unruptured cerebral aneurysm

Exclusion Criteria:

* Patients not able to read, or understand the consent form
* Ethnicity, other than Korean population
* Patients refusal
* Patients not to perform total intravenous anesthesia
* Patients currently taking psychiatric medication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean adult population undergoing propofol based total intravenous anesthesia for clipping of unruptured cerebral aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Time of eye opening after stopping propofol infusion | Within one hour
  When operation is finished, investigator will stop the intravenous infusion of propofol. Investigators will measure the time from when propofol infusion is stopped until eye opening and extubation, respectively. The measurement will be established within about one hour from end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iohom G, Ni Chonghaile M, O'Brien JK, Cunningham AJ, Fitzgerald DF, Shields DC. An investigation of potential genetic determinants of propofol requirements and recovery from anaesthesia. Eur J Anaesthesiol. 2007 Nov;24(11):912-9. doi: 10.1017/S0265021507000476. Epub 2007 Jun 7. PMID 17555608